CLINICAL TRIAL: NCT02121028
Title: Mechanisms of Early Recurrence in Intracranial Atherosclerotic Disease
Acronym: MyRIAD
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: University of California, Los Angeles (Other); Northwestern University (Other); Emory University (Other); Baystate Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jose Romano, MD, Professor of Clinical Neurology, University of Miami
Other Study IDs: 20140056; 1R01NS084288-01A1 (NIH)
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Intracranial Vascular Disorders
Keywords: Intracranial Atherosclerotic Disease; Stroke; Transient Ischemic Attack; Imaging
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracranial Atherosclerotic Disease, Stroke/TIA: Stroke/TIA due to high grade IAD ≤21 days from symptom onset.

SUMMARY:
The objective of this study is to determine the mechanisms of stroke in patients with Intracranial Atherosclerotic Disease (IAD) by specifically evaluating limitations of antegrade flow through the stenotic artery, distal tissue perfusion to the affected territory, and artery-to-artery embolism. The hypothesis is that non-invasive imaging biomarkers that stratify stroke risk and distinguish mechanisms of IAD. This prospective multicenter study will enroll 175 patients with recently symptomatic high-grade IAD. Patients will be studied within 21 days of the index event (allowing appropriate time to arrange for diverse imaging modalities), with the following advanced neuroimaging techniques to elucidate mechanisms of recurrent ischemia:

* Quantitative magnetic resonance imaging (QMRA) to assess volumetric flow rate through the stenotic artery.
* Magnetic resonance perfusion weighted imaging (PWI-MRI) to determine distal tissue perfusion.
* Vasomotor reactivity by Transcranial Doppler using the breath-holding technique (BHI-TCD) to assess compensatory flow characteristics to the territory distal to the affected artery;
* Transcranial Doppler with embolic signal monitoring to evaluate artery-to-artery embolism that reflects plaque instability.

Patients will receive standardized medical management and its effectiveness on blood pressure, lipid, and glycemic control will be monitored.

The primary outcome is recurrent stroke in the territory of the stenotic artery during a 1-year follow-up period; secondary outcomes are: a) new asymptomatic ischemic lesions on MRI in the distribution of the stenotic artery at 6-8 weeks, and b) transient ischemic attack (TIA) in the distribution of the stenotic artery during a 1-year follow-up period.

Patients will be recruited at various sites that will be trained and certified on the imaging techniques employed. Raw imaging data will be interpreted centrally.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke defined as symptoms lasting >24 hours and associated with imaging evidence of acute ischemia in the distribution of the stenotic vessel on CT or MRI.
2. Eligible TIA defined as transient neurological symptoms lasting <24 hours, need to be:

   1. accompanied by DWI abnormalities in the distribution of the stenotic artery; or
   2. multiple (≥2), stereotyped events associated with unequivocal ischemic symptoms (weakness, aphasia), and attributed to the symptomatic artery.
3. IAD should involve the intracranial carotid, middle cerebral, intracranial vertebral or basilar arteries.
4. Stenosis 50-99% quantified by digital subtraction angiography (DSA), CT angiography-CTA or MR angiography-MRA tests. DSA is not required but will be used if obtained as part of clinical care.

   The criteria for 50-99% are:
   1. CTA or DSA: measured 50-99% stenosis by WASID criteria (percent stenosis = (1-[diameter stenosis/diameter normal]) x 100%.
   2. MRA: measured 50-99% stenosis or presence of a flow gap.
5. Age >30; those 30-49 years of age must also have the presence of established atherosclerotic disease in another vascular bed (coronary, extracranial carotid, peripheral) or the presence of 2 or more risk factors (hypertension, diabetes mellitus, hyperlipidemia, tobacco abuse within the last 2 years).
6. Enrollment within 21 days of symptom onset and completion of study imaging tests within 21 days of index event (stroke or TIA).
7. Provide informed consent for participation in the study.

Exclusion Criteria:

1. Other cause for stroke: atrial fibrillation, acute anterior wall ST-elevation myocardial infarction <30days, mitral stenosis, mechanical valve, intracardiac thrombus or vegetation, dilated cardiomyopathy or ejection fraction <30%, proximal extracranial carotid or vertebral stenosis >50%.
2. Contraindications to MRI, including MR-incompatible metallic implants, implanted electronic devices, other potentially mobile ferromagnetic material, pregnancy (women in fertile age should have a negative pregnancy test), lactation, morbid obesity, and severe claustrophobia.
3. Renal impairment defined as either a creatinine level >1.5 mg/dL or a glomerular filtration rate (GFR) <30 mL/min/1.73 m2.
4. Known allergy to gadolinium.
5. Unable to obtain informed consent by patient or legally authorized representative.
6. Severe behavioral or social problems that may interfere with the conduct of the study.
7. In the investigator's opinion, patient unlikely return for follow up visit and to complete the study.
8. Participation in a drug or device clinical trial within the last 30 days.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have a recent stroke or TIA due to intracranial Atherosclerotic Disease (IAD) of 50-99% .
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrent stroke in the territory of the symptomatic artery | 1 year
  Time to ischemic stroke in the territory of the symptomatic artery. Stroke is ascertained by the site neurologist and defined as new or worsening symptoms lasting >24 hours and associated with imaging evidence of ischemia on CT or MRI in the distribution of the stenotic artery.

SECONDARY OUTCOMES:
TIA in the territory of the stenotic artery | 1 year
  TIA in the territory of the stenotic artery is defined as transient neurological symptoms lasting <24 hours and clearly related to the stenotic artery as per a neurologist.
Silent infarcts in the distribution of the stenotic artery | 6-8 weeks
  Silent infarcts will be assessed by comparing the DWI and FLAIR sequences at baseline and at 6-8 weeks. Silent infarcts are defined as new discrete lesions not apparent in the baseline images that are in the distribution of the stenotic artery, in the absence of the primary endpoint.

OTHER OUTCOMES:
Risk of combined microembolic signals and impaired vasomotor reactivity. | 1 year
  Assess the interaction of the presence of micro embolic signals, assessed by TCD and a marker of plaque emboligenecity, and impaired vasomotor reactivity, assessed by TCD and a marker of collateral flow limitation, in increasing the risk of recurrent stroke in the territory of the target artery.
Risk of combined poor ante grade flow and poor distal tissue perfusion. | 1 year
  Assess the Interaction between two mechanisms of cerebral ischemia, poor antegrade flow assessed by quantitative MRA as a marker of flow across a stenotic arterial segment, and poor tissue perfusion assessed by perfusion MRI and representative of distal territorial perfusion, in the risk of recurrent stroke in the territory of the stenotic artery.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Romano, MD, Principal Investigator — University of Miami; Shyam Prabhakaran, MD, Principal Investigator — University of Chicago; David S Liebeskind, MD, Principal Investigator — University of California, Los Angeles
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Northwestern University Department of Radiology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prabhakaran S, Liebeskind DS, Cotsonis G, Nizam A, Feldmann E, Sangha RS, Campo-Bustillo I, Romano JG; MYRIAD Investigators. Predictors of Early Infarct Recurrence in Patients With Symptomatic Intracranial Atherosclerotic Disease. Stroke. 2021 Jun;52(6):1961-1966. doi: 10.1161/STROKEAHA.120.032676. Epub 2021 Apr 19. PMID 33866818
- [Derived] Romano JG, Prabhakaran S, Nizam A, Feldmann E, Sangha R, Cotsonis G, Campo-Bustillo I, Koch S, Rundek T, Chimowitz MI, Liebeskind DS; MyRIAD Investigators. Infarct Recurrence in Intracranial Atherosclerosis: Results from the MyRIAD Study. J Stroke Cerebrovasc Dis. 2021 Feb;30(2):105504. doi: 10.1016/j.jstrokecerebrovasdis.2020.105504. Epub 2020 Dec 1. PMID 33276302